CLINICAL TRIAL: NCT07138937
Title: Efficiency of Sonic Activation During Root Canal Treatment of Primary Molars on Postoperative Pain and Facial Expressions of Children Using Artificial Intelligence
Brief Title: Efficiency of Sonic Activation During Root Canal Treatment of Primary Molars on Postoperative Pain and Facial Expressions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 728/2024
Record Dates: First submitted 2025-08-02; First posted 2025-08-24 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Root Canal Treatment in Children Primary Molars; Postoperative Pain; Facial Expressions; Facial Emotions; Artificial Intelligence Mobile Application; Sonic Activation
Keywords: Sonic activation; Postoperative pain; Primary molars; AI applications; Facial emotions
MeSH Terms: conditions — Pain, Postoperative; Facial Expression

STUDY DESIGN:
Intervention Model Description: A comparative, randomized, prospective clinical trial to evaluate the efficacy of sonic activation versus no activation by comparing the pain scale and facial expressions following root canal treatment in primary molars.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sonic activation of irrigation (Active Comparator): Sonic activation of irrigation with Eddy system
  Interventions: Procedure: Root canal treatment in primary molars with irreversible pulpitis; Device: EDDY system for sonic activation of irrigation
- No activation (Placebo Comparator): Irrigation with side-vented needle without activation
  Interventions: Procedure: Root canal treatment in primary molars with irreversible pulpitis; Device: side-vented needle

INTERVENTIONS:
Procedure: Root canal treatment in primary molars with irreversible pulpitis — Root canal treatment in primary molars with irreversible pulpitis followed by coronal restoration with stainless-steel crowns in a single visit.
Device: EDDY system for sonic activation of irrigation — sonic activation of irrigation with EDDY system during root canal treatment in primary molars
  Arms: Sonic activation of irrigation
Device: side-vented needle — conventional irrigation with side-vented needle without activation during root canal treatment in primary molars
  Arms: No activation

SUMMARY:
This study was conducted to evaluate the efficiency of sonic activation of 5%sodium hypochlorite during root canal treatment of primary molars on postoperative pain and facial expressions. In addition to comparing between the Five-face pain scale and AI Emotion Detector mobile application in postoperative pain assessment.

DETAILED DESCRIPTION:
The current study addresses an important gap in research, as the impact of sonic activation of irrigation on postoperative pain in children and the validity of artificial intelligence mobile application in detecting facial expressions following root canal treatment as not been well explored.

ELIGIBILITY:
Inclusion Criteria:

1. Children's age range 5-8 years. Boys and girls will be included.
2. Children with positive or definitely positive behavior on the Frankl's behavior rating scale (rating 3 or 4 on the scale).
3. Children with at least one primary molar with irreversible pulpitis and symptomatic apical periodontitis confirmed using periapical radiographs, percussion, and cold test.
4. Children having teeth with two-thirds of each root remaining.
5. Children with a moderate to very severe (2-4) pain score according to five-face pain scale in only one tooth within the 24-h period before the procedure.
6. Children with no allergy to Ibuprofen.

Exclusion Criteria:

1. Teeth with pathological root resorption.
2. Teeth with mobility greater than 1st-degree mobility.
3. Children who received analgesics and/or antibiotics in the last 12 h before root canal treatment

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Five-Face Pain Scale Score | 8 ,24,48,72 hours, and after 1week post-operative
  Postoperative pain is assessed using the Five-Face Pain Scale (range: 0 = no pain to 4= worst pain; lower scores indicate less pain).
  Unit of Measure: Scale units (0-4)
facial expressions analysis | 8 ,24,48,72 hours, and after 1week post-operative
  facial expressions of the patients are assessed from their photographs and analyzed by the AI Emotion Detector mobile application.
  Unit of Measure: Percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Abdelhamid El-Baz, Professor of Pedodontics, Study Chair — Faculty of dentisrty, Suez Canal University
Locations (1):
- Faculty of Dentistry Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to patient confidentiality restrictions.